CLINICAL TRIAL: NCT04505098
Title: A Pragmatic Randomized Trial of Icosapent Ethyl for High-Cardiovascular Risk Adults (MITIGATE)
Brief Title: A Pragmatic Randomized Trial of Icosapent Ethyl for High-Cardiovascular Risk Adults
Acronym: MITIGATE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was suspended by the IRB of record and subsequently terminated
Sponsor: Kaiser Permanente (Other)
Collaborators: Amarin Corporation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1597940
Record Dates: First submitted 2020-08-05; First posted 2020-08-10 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Covid19; Atherosclerosis; Cardiovascular Diseases; Upper Respiratory Tract Infections
MeSH Terms: conditions — COVID-19; Atherosclerosis; Cardiovascular Diseases; Respiratory Tract Infections | interventions — eicosapentaenoic acid ethyl ester

STUDY DESIGN:
Intervention Model Description: Pragmatic randomized clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator)
  Interventions: Drug: Icosapent ethyl
- Usual Care (No Intervention)

INTERVENTIONS:
Drug: Icosapent ethyl — 2 g by mouth twice daily for at least 6 months
  Other Names: Vascepa
  Arms: Intervention

SUMMARY:
MITIGATE is a prospective, open-label, parallel-group, randomized, pragmatic clinical trial. The MITIGATE Study has been designed to evaluate the real-world clinical effectiveness of pre-treatment with icosapent ethyl (IPE), also known as Vascepa®, compared to usual standard of care to prevent and reduce the sequelae of laboratory-confirmed viral upper respiratory infection (URI)-related (i.e., COVID-19, influenza, and other known viral respiratory pathogens) morbidity and mortality in a high-risk cohort of adults with established atherosclerotic cardiovascular disease (ASCVD).

DETAILED DESCRIPTION:
For the MITIGATE study, eligible members receiving care within Kaiser Permanente Northern California (KPNC) will be identified and screened electronically in a 1:10 intervention to control allocation (i.e., IPE vs. usual care) stratified by age and pre-existing respiratory status. Patients randomly assigned and enrolled into the intervention arm will be asked to take IPE (2 grams by mouth twice daily) for a minimum of 6 months and until study completion. Patients assigned to the control arm (i.e., usual care) will be passively followed only electronically via the electronic health record (EHR).

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent (for the intervention arm only)
* No prior history of confirmed COVID-19 (i.e., based on a positive FDA-approved assay for SARS-CoV-2 and no documented FDA-approved serological test results for antibodies to SARS-CoV-2 found in health system databases)
* Established ASCVD (i.e., defined as prior myocardial infarction, percutaneous coronary intervention, coronary artery bypass surgery, ischemic stroke, and/or peripheral artery disease)
* At least 12 months of continuous health plan membership and prescription drug benefit prior to enrollment
* A registered e-mail address with the health care delivery system in order to facilitate obtaining electronic consent for study participation

Exclusion Criteria:

* Receipt of IPE on or within 12 months before the day of enrollment
* Known hypersensitivity to IPE, fish, and/or shellfish
* Documented use of any omega-3 fatty acid medications or dietary supplements containing omega-3 fatty acids in the EHR
* Women who are pregnant or planning to become pregnant
* Hospitalization for myocardial infarction and/or elective percutaneous coronary intervention within the past 1 month
* Currently receiving triple anti-thrombotic therapy
* Stage D heart failure
* Severe liver disease
* End-stage renal disease requiring chronic dialysis or estimated glomerular filtration rate <15 mL/min/1.73 m2
* Metastatic cancer and/or receiving active systemic chemotherapy
* Institutionalized and/or receiving palliative care

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39600 (Actual)
Dates: Start 2020-08-07 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Rate of confirmed viral URIs | 0-12 months
  Confirmed viral URIs (i.e., including recurrent events) (i.e., COVID-19, influenza, and other known viral respiratory pathogens) based on laboratory testing (i.e., FDA or locally-approved testing modalities)

SECONDARY OUTCOMES:
Percentage of patients with moderate or severe confirmed viral URIs | 0-12 months
  Confirmed viral URIs (i.e., including recurrent events) (i.e., COVID-19, influenza, and other known viral respiratory pathogens) based on laboratory testing (i.e., FDA or locally-approved testing modalities) with an oxygen saturation <94% on room air and/or requiring any form of supplemental oxygen.
Worst clinical status due to a confirmed viral URI | 0-12 months
  At any point in time based on a 7-point ordinal scale (i.e., 1 = death, 2 = mechanically ventilated/extracorporeal membrane oxygenation, 3 = high flow supplemental oxygen, 4 = low flow supplemental oxygen, 5 = hospitalized with no supplemental oxygen requirements, 6 = urgent care or emergency department visit not leading to hospitalization, and 7 = no relevant clinical encounters)

OTHER OUTCOMES:
Percentage of participants who die due to any cause | 0-12 months
Percentage of participants experiencing a major adverse cardiovascular event | 0-12 months
  Death due to any cause, hospitalization for myocardial infarction, or hospitalization for ischemic stroke
Percentage of participants experiencing an expanded major adverse cardiovascular event | 0-12 months
  Major adverse cardiovascular events, hospitalization for acute coronary syndrome, and coronary revascularization (i.e., percutaneous coronary intervention and/or coronary artery bypass graft)
Percentage of participants who are hospitalized for heart failure | 0-12 months
Percentage of participants who are hospitalized for any reason | 0-12 months
Percentage of participants who have an emergency department visit for any reason | 0-12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Research, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: No